CLINICAL TRIAL: NCT01985165
Title: A Multicenter，Open-label Phase Ⅳ Trial of Imrecoxib in Treatment of Knee Osteoarthritis
Brief Title: A Phase 4 Study of Imrecoxib in Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRARXB00434
Record Dates: First submitted 2013-11-01; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Imrecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imrecoxib (Experimental): 0.1g,BID,po
  Interventions: Drug: Imrecoxib

INTERVENTIONS:
Drug: Imrecoxib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Imrecoxib in the treatment of patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Aged form 18 years to 75 years old
* Diagnosed with osteoarthritis of the knee according to the American College of Rheumatology
* Functional capacity class of Ⅰ-Ⅲ

Exclusion Criteria:

* Unstable angina
* History of myocardial infarction within the last 6 months
* Stroke in the 6 months before screening
* New York Heart Association class Ⅲ-Ⅳ congestive heart-failure
* Systolic blood pressure>180mmHg,and/or Diastolic blood pressure>100mmHg
* Peptic ulcer
* Known contraindications to non-steroidal anti-inflammatory drug（NSAID）
* Received aspirin within 3 days of baseline visit
* Aspirin dosage>150mg/d
* Known to be Allergic to sulfa and COX-2 inhibitors
* Pregnancy or lactation
* Glutamic-oxaloacetic transaminase and/or glutamic-pyruvic transaminase>2 times upper limit of normal
* Blood urine nitrogen>1.5 times upper limit of normal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Patient's Assessment of Arthritis Pain, according to Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)3.0 | Baseline to Week 24
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Fengchun Zhang, Professor, Principal Investigator — Peking Union Medical College Hospita
Locations (19):
- China (19):
  - The Second Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Tongji Hospital, Wuhan, Hubei
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Qianfoshan Hospital Affiliated to Shandong University, Jinan, Shandong
  - The Second Hospital of Shangdong University, Jinan, Shandong
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital, Taizhou, Zhejiang
  - BeijingChao-YangHospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Hospital of the Ministry of Health, Beijing
  - Peking Union Medical College Hospita, Beijing
  - Peking University Third Hospital, Beijing
  - Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing
  - Tianjin First Center Hospital, Tianjin